CLINICAL TRIAL: NCT03278496
Title: Recovery Housing and Drug Abuse Treatment Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DA13003
Record Dates: First submitted 2014-03-28; First posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Mental and Behavioral Disorders Due to Use of Cocaine: Harmful Use; Opiate Addiction
Keywords: addiction; substance abuse treatment; aftercare; outpatient counseling; opiates; cocaine
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Recovery housing plus counseling (Experimental): Intensive counseling in a 5-day per week program plus abstinence-contingent rent payment in a community recovery house. Intervention lasts 12 weeks with follow-up at 12 and 24 weeks post treatment entry.
  Interventions: Behavioral: Recovery Housing plus Counseling
- Recovery Housing only (Experimental): Abstinence-contingent payment for recovery housing rent in absence of any formal counseling. Intervention lasts 12 weeks with follow-up at 12 and 24 weeks post treatment entry.
  Interventions: Behavioral: Recovery Housing Only
- Usual Care Referral (Active Comparator): Participants receive referral resources for community substance abuse counseling and recovery housing but no formal treatment or help with rent payments. All participate in follow-up data collection.
  Interventions: Behavioral: Usual Care Referral

INTERVENTIONS:
Behavioral: Recovery Housing plus Counseling — Participants receive 3 months of abstinence-contingent program-supported rent payment in community recovery housing. They also receive intensive outpatient counseling (both individual and group) focused on relapse prevention skills training, goal setting, employment seeking and recreational activities.
  Arms: Recovery housing plus counseling
Behavioral: Usual Care Referral — Participants are referred to an outpatient program of their choosing with an appointment made for them.
  Arms: Usual Care Referral
Behavioral: Recovery Housing Only — Participant may receive up to 3 months of abstinence-contingent rent payment in community recovery housing but is not invited to participate in intensive counseling.
  Arms: Recovery Housing only

SUMMARY:
Reinforcement-Based Therapy (RBT) is an intensive outpatient substance abuse treatment that includes relapse prevention skills training, goal setting, help with finding employment and abstinence-contingent rent payment for recovery housing in the community. It is meant to provide motivation for continued abstinence while enhancing social stability. In this study, treatment was offered to inner city opiate and cocaine users immediately following a brief medically-supported residential detoxification. Previous research had shown that RBT produces 3- month outcomes superior to those for patients who are referred to outpatient treatment in the community. The present study compared outcomes for patients (N = 243) randomly assigned to receive abstinence-contingent recovery housing with (full RBT) or without additional intensive counseling or to receive usual care referral to outpatient treatment following detoxification. Outcomes were similar at 3- and 6-month follow-ups for those who received recovery housing with (full RBT) and without additional counseling and both these treatments were superior to usual care referral. Study findings support the efficacy of post-detoxification recovery housing with or without counseling for opiate and cocaine users.

DETAILED DESCRIPTION:
Aims To conduct a randomized, controlled trial of abstinence-contingent recovery housing delivered with or without intensive day treatment among individuals exiting residential opioid detoxification.

Design Random assignment to one of three conditions: recovery housing alone (RH), abstinence-contingent recovery housing with reinforcement-based treatment RBT (RH + RBT) or usual care (UC). RH and RH + RBT participants received 12 weeks of paid recovery housing contingent upon drug abstinence. RH + RBT participants also received 26 weeks of RBT, initiated concurrently with recovery housing. Assessments were conducted at 1, 3 and 6 months after treatment enrollment.

Setting Out-patient drug-free substance abuse treatment program in Baltimore, Maryland.

Participants Patients (n = 243) who completed medication-assisted opioid detoxification.

Measurements Primary outcome was drug abstinence (opioid- and cocaine-negative urine and no self-reported opioid or cocaine use in the previous 30 days). Secondary outcomes included abstinence at all time-points (1, 3 and 6 months), days in recovery housing and employment.

ELIGIBILITY:
Inclusion Criteria:

* completes residential detoxification for use of opiates and/or cocaine
* willing to go to outpatient aftercare
* agrees to random assignment; signs informed consent

Exclusion Criteria:

* moving out of town
* primary substance use does not include opiates or cocaine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 243 (Actual)
Dates: Start 2001-04; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
abstinence from opiates and cocaine | 6 months post randomization
  Free in the community plus self report of no drug use in past 30 days verified with negative urine screen.

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Stitzer, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Result] Tuten M, DeFulio A, Jones HE, Stitzer M. Abstinence-contingent recovery housing and reinforcement-based treatment following opioid detoxification. Addiction. 2012 May;107(5):973-82. doi: 10.1111/j.1360-0443.2011.03750.x. Epub 2012 Feb 28. PMID 22151478